CLINICAL TRIAL: NCT04945538
Title: Quantification and Determinants of Occupational Xray Scatter Radiation Exposure of Operators and Assistants During Coronary Procedures - The Occupational SCAtter Radiation Registry
Brief Title: Scatter Radiation Exposure During Coronary Procedures - The Occupational SCAtter Radiation Registry
Acronym: OSCAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Mathias Brandt, MD, Senior Physician, Principal Investigator, Paracelsus Medical University
Other Study IDs: ParacelsusMU
Record Dates: First submitted 2021-06-21; First posted 2021-06-30 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Scatter radiation exposure measurement — Scatter radiation exposure of the operator and sterile assistant is recorded with digital live dosimeters at 3 locations of the operator (frontal head at eye level, left lateral head, below the left shoulder) and at 2 locations of the sterile assistant (left neck and below the left shoulder)

SUMMARY:
During diagnostic and interventional coronary procedures scatter radiation exposure is recorded with live-dosimeters at pre-specified anatomic regions of operators and sterile assistants. Scatter radiation data is correlated with detailed Xray exposure data and technical details of the procedure.

The purpose of the registry is:

1. to establish scatter radiation reference values based on a large number of representative cath-lab procedures
2. to identify technical and clinical factors predisposing for high scatter radiation exposure,
3. to evaluate advanced radiation protection devices in clinical routine.

DETAILED DESCRIPTION:
Patients scheduled for diagnostic or interventional coronary procedures provide written informed consent for participating in the observational OSCAR Registry. During the corresponding procedures, scatter radiation exposure of operators and sterile assistants is recorded using Unfors RaySafe i3 digital live dosimeters (Unfors RaySafe AB, Billdal, Sweden) at 3 locations of the operator (1-frontal head at eye level, 2-left lateral head, 3-below the left shoulder) and at 2 locations of the sterile assistant (1-left neck and 2-below the left shoulder).

Raw data is collected in a central database and correlated with patient properties (age, BMI) and detailed Xray exposure data:

* Total dose-area product (DAP, unit of measure: Gy*cm2)
* Number of Xray image series
* Number of Images
* Radiation duration (Unit of measure: Seconds)
* Air kinetic energy released per unit mass (Kerma) Technical details of the procedure
* Access site,
* Clinical setting: acute or elective
* Number of catheters used during procedure
* Number of guidewires used during procedure
* Number of stents implanted during procedure
* Cumulative stent length (Unit of measure: mm)
* Use of rotational imaging
* Use of intracoronary pressure-wire
* Use of optical coherence tomography (OCT)
* Presence of bypass-vessels
* Any occurrence of complications

The purpose of the trial is to establish a large foundation of intra-procedural scatter radiation data from representative coronary procedures procedures enabling our group to

1. Establish scatter radiation reference values based on a large number of representative cath-lab procedures
2. Identify technical and clinical factors predisposing for high staff scatter radiation exposure
3. Evaluate advanced radiation protection devices in clinical routine.

This includes:

* Additional ceiling-suspended lead-shielding
* Ceiling-suspended radiation protection devices like the "Zero-Gravity"-System (TIDI Medical Products, Neenah, WI, USA)
* Patient lead-covers.

The study was submitted to and approved by the federal Ethics Committee Salzburg (reference number ECS 1069/2021).

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for coronary angiography
* Diagnostic procedure and PCI
* Acute and elective procedures
* Standard percutaneous coronary interventions (PCI) interventions
* Chronic total occlusion (CTO) interventions
* Set of at least 4 personal digital live dosimeters (PDL) worn by operator and sterile assistant for the entire duration of the procedure
* Staff (operators and assistants) instructed on PDL positioning prior to procedure

Exclusion Criteria:

* Less than 4 PDL present during the procedure
* Incomplete data recording by at least 1 PDL
* PDL data cannot be unambiguously assigned to a specific procedure or a specific anatomical recording site
* Exchange of operator or assistant during procedure without transfer of all PDL

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Two study populations have to be considered separately:
  1. PDL Recordings:
     Study population: Interventional cardiologists regularly assigned to our Cath-labs working at the cath-lab table during the majority of their assignment.
  2. Coronary procedures during which data is recorded:
  Study population: Patients with clinical indication for diagnostic or interventional coronary procedures, representing the classic cardiologic patient population with suspected or known coronary artery disease, acute coronary syndrome or heart valve dysfunction.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2025-08-08 (Estimated); Study Completion 2025-09-08 (Estimated)

PRIMARY OUTCOMES:
Intra-procedural Xray scatter radiation exposure (µSv) | Duration of procedure
  Xray scatter radiation dose recorded by 5 personal live dosimeters (3 allocated to the operator, 2 allocated to the sterile assistant).

CONTACTS AND LOCATIONS:
Locations (1):
- Paracelsus Medical University, Clinic II of Internal Medicine, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brandt M, Prinz E, Schernthaner C, Kraus J, Wintersteller W, Hammerer M, Strohmer B, Lichtenauer M, Motloch L, Hoppe UC, Nairz O. Advanced Radiation Protection in PCI and Diagnostic Procedures With a Ceiling-Suspended Radiation Protection System-Data From the OSCAR Registry. J Am Coll Cardiol 2021; 78 (19_Supplement_S): B63-B64
- See also: Austrian Society of Cardiology 2021 Poster — http://stage-atcardio.multimedium.at/storage/app/media/Jahrestagung/POSTER/Interventionelle%20Kardiologie/Brandt%20.pdf